CLINICAL TRIAL: NCT04569968
Title: Effect of Expiratory Muscle Training on Stomatognathic System in Patients With Stroke
Brief Title: Expiratory Muscle Training in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAIBU-FTR-ÖD-01
Record Dates: First submitted 2020-08-26; First posted 2020-09-30 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Mastication Disorder; Temporomandibular Disorders; Dysphagia; Stomatognathic Diseases
Keywords: Stroke; Mastication; Dysphagia; Temporomandibular joint
MeSH Terms: conditions — Stroke; Temporomandibular Joint Disorders; Deglutition Disorders; Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Two groups as an intervention and control.
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be performed by an another investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory muscle training group (Experimental): Daily expiratory muscle training for four weeks will be applied.
  Interventions: Other: Expiratory muscle training
- Control group (No Intervention): Nothing will be applied except for the hospital conventional physiotherapy program.

INTERVENTIONS:
Other: Expiratory muscle training — For training group first maximum expiratory pressure measurement will be assessed with portable expiratory measurement device. Measurement will be taken while the patient in a sitting position. Three measurement values with 5% variation will be taken an average of these values recorded as a maximum expiratory pressure of the patient. After the maximum expiratory pressure of the patient is measured 50% percent of the related value will be set on the expiratory muscle trainer. Then patient will be informed about how to use the trainer. Trainer will be used daily for four weeks with 50 repetitions. At the end of every week pressures will be measured again for re-calibration of the trainer.
  Arms: Expiratory muscle training group

SUMMARY:
Stroke affects the vital activities of daily living such as breathing and swallowing. After stroke excursion of the diaphragm reduces about 50%, and also the maximum expiratory pressure of the individual 50% or higher. Dysphagia occurs in 29% to 45% of the acute stroke cases.

DETAILED DESCRIPTION:
As a third leading cause of death and one of the major causes of disability, stroke still maintain its bad reputation in worldwide. Stroke owes its fame on wide range of symptoms mostly the musculoskeletal system symptoms such as spasticity, equilibrium and gait problems. Although mentioned symptoms keep their popularity devious two dysfunction caused by stroke; stomatognathic system dysfunction and respiratory dysfunction appears to change this equation. Considering the high incidence of dysphagia and the reduced cardiopulmonary capacity of the stroke patients, it seems inevitable. From this perspective aim of this study is to assess the effect of expiratory muscle training on the stomatognathic system in patients with stroke and as mentioned aid to shatter the mentioned equation.

ELIGIBILITY:
Inclusion Criteria:

* Mini mental score is 24 or higher
* 55 years of age or higher
* Currently not taking respiratory muscle training
* Fonseca Questionnaire score is 20 or higher
* Onset of stroke is between 3 months and 5 years

Exclusion Criteria:

* Developed dysphagia caused by other diseases rather than stroke
* Repetitive stroke story
* Cancer in head and neck region
* Abdominal or thoracic surgery story
* Existence of neurodegenerative disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Dursun, MSc, Principal Investigator — Bolu Abant İzzet Baysal University; Tamer Çankaya, PhD, Principal Investigator — Bolu Abant İzzet Baysal University; Erdal Dilekçi, MD, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (2):
- Turkey (Türkiye) (2):
  - İzzet Baysal Physical Therapy and Rehabilitation Education and Research Hospital, Bolu
  - Bolu Abant İzzet Baysal University, Bolu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Similowski T, Catala M, Rancurel G, Derenne JP. Impairment of central motor conduction to the diaphragm in stroke. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):436-41. doi: 10.1164/ajrccm.154.2.8756819.
- [Background] Finestone HM, Greene-Finestone LS, Wilson ES, Teasell RW. Malnutrition in stroke patients on the rehabilitation service and at follow-up: prevalence and predictors. Arch Phys Med Rehabil. 1995 Apr;76(4):310-6. doi: 10.1016/s0003-9993(95)80655-5. PMID 7717830
- [Background] Khedr EM, El Shinawy O, Khedr T, Abdel aziz ali Y, Awad EM. Assessment of corticodiaphragmatic pathway and pulmonary function in acute ischemic stroke patients. Eur J Neurol. 2000 Sep;7(5):509-16. doi: 10.1046/j.1468-1331.2000.00104.x. PMID 11054135
- [Background] Messaggi-Sartor M, Guillen-Sola A, Depolo M, Duarte E, Rodriguez DA, Barrera MC, Barreiro E, Escalada F, Orozco-Levi M, Marco E. Inspiratory and expiratory muscle training in subacute stroke: A randomized clinical trial. Neurology. 2015 Aug 18;85(7):564-72. doi: 10.1212/WNL.0000000000001827. Epub 2015 Jul 15. PMID 26180145
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Yelnik AP, Le Breton F, Colle FM, Bonan IV, Hugeron C, Egal V, Lebomin E, Regnaux JP, Perennou D, Vicaut E. Rehabilitation of balance after stroke with multisensorial training: a single-blind randomized controlled study. Neurorehabil Neural Repair. 2008 Sep-Oct;22(5):468-76. doi: 10.1177/1545968308315996. PMID 18780882
- [Background] Sommerfeld DK, Eek EU, Svensson AK, Holmqvist LW, von Arbin MH. Spasticity after stroke: its occurrence and association with motor impairments and activity limitations. Stroke. 2004 Jan;35(1):134-9. doi: 10.1161/01.STR.0000105386.05173.5E. Epub 2003 Dec 18. PMID 14684785
- [Background] Dursun O, Cankaya T. Assessment of Temporomandibular Joint Dysfunction in Patients with Stroke. J Stroke Cerebrovasc Dis. 2018 Aug;27(8):2141-2146. doi: 10.1016/j.jstrokecerebrovasdis.2018.03.007. Epub 2018 Apr 9. PMID 29650380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from İzzet Baysal Physical Therapy Education and Research Hospital between 18.08.2020 and 06.09.2021.
Pre-assignment Details: Patients who had the following situations were excluded from the study; stroke onset of time higher than 3 months, hemorrhagic stroke, cooperation problem, age of 64 or younger, denial of participation to the study, head and/or neck surgery existence, discharge, free of temporomandibular joint dysfunction, existence of infection, incisor and/or canin tooth absence, quarantine, insufficient mastication.
Groups:
- Expiratory Muscle Training Group: Daily expiratory muscle training for three weeks with 50 repetition was applied to the experimental group.
- Control Group: Nothing applied except for the hospital conventional physiotherapy program.
Period: Overall Study
Arm/Group | Expiratory Muscle Training Group | Control Group
Started | 86 | 60
Completed | 15 | 16
Not Completed | 71 | 44
Not completed — Lost to Follow-up | 2 | 5
Not completed — Story of head and/or neck surgery | 2 | 2
Not completed — Time of stroke onset | 8 | 7
Not completed — Type of strokr | 12 | 8
Not completed — Cooperation | 8 | 8
Not completed — Age interval | 17 | 6
Not completed — Denial of participation to the study | 0 | 3
Not completed — Free of temporomandibular joint dysfunction | 4 | 2
Not completed — Lack of incisor and/or canin tooth | 5 | 3
Not completed — Quarantine | 1 | 0
Not completed — Previous recruitment to the expiratory muscle training | 2 | 0
Not completed — Repetitive stroke | 8 | 0
Not completed — Insufficient mastication | 1 | 0
Not completed — Infection | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Expiratory Muscle Training Group | Control Group | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 5 | 9 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 11 | 7 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Masticatory Performance
Description: To assess masticatory performance of the patients, patients will be asked to chew 3 gr of peanuts with 20 chewing stroke and then spit on a sieve with 10 mesh and 1700 µm width. Then the residue will be collected and put into the centrifuge tube. After that residue will be centrifuged for 3 minutes with 1500 rpm. Same procedure will be used for the sieved content. Then this two values will be divided and recorded as a percentage for the calculation masticatory performance index.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Mean (Standard Deviation); unit: percentage of masticated peanuts
Groups:
- Expiratory Muscle Training Group: Daily expiratory muscle training for three weeks will be applied.
  Expiratory muscle training: For training group first maximum expiratory pressure measurement will be assessed with portable expiratory measurement device. Measurement will be taken while the patient in a sitting position. Three measurement values with 5% variation will be taken an average of these values recorded as a maximum expiratory pressure of the patient. After the maximum expiratory pressure of the patient is measured 50% percent of the related value will be set on the expiratory muscle trainer. Then patient will be informed about how to use the trainer. Trainer will be used daily for four weeks with 50 repetitions. At the end of every week pressures will be measured again for re-calibration of the trainer.
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
percentage of masticated peanuts
  First measurement | 24 (18) | 13 (7)
  Last measurement | 25 (17) | 16 (10)

2. Primary Outcome: Change in Temporomandibular Range of Motion Measurement
Description: Mandibular depression, protrusion and bilateral lateral deviation of the patients will be performed by a digital caliper. All measurements will be taken while the patients are seated with their head supported. Digital caliper will be positioned in central incisors for the mandibular depression and the protrusion. For lateral deviation first upper central incisor location in relation to the lower central incisor will be drawn by a biocompatible pen then measurement will be performed. After that, a second drawing made. Then the horizontal distance between these two points will be measured for the lateral deviation range of motion. Reference values for mandibular depression, protrusion and the lateral deviation are as follows: 40 mm, 6 mm, and 8 mm.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Mean (Standard Deviation); unit: milimeter
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
milimeter
  Mandibular depression first measurement | 39.55 (6.42) | 41.48 (7.40)
  Mandibular depression last measurement | 41.90 (6.71) | 41.09 (7.10)
  Left lateral deviation first measurement | 7.61 (2.97) | 5.25 (2.33)
  Left lateral deviation last measurement | 6.84 (1.92) | 5.49 (1.98)
  Right lateral deviation first measurement | 7.44 (2.04) | 5.54 (2.49)
  Right lateral deviation last measurement | 8.09 (2.34) | 5.61 (2.15)
  Protrusion first measurement | 5.28 (1.61) | 4.17 (1.83)
  Protrusion last measurement | 5.56 (1.18) | 4.62 (2.21)

3. Primary Outcome: Change in General Oral Health Assessment Index
Description: Oral health of the patients will be assessed with general oral health assessment index. Index consists of twelve questions. Answers of these twelve questions makes up the total score. Minimum and maximum scores of the index are 12 and 60 points. Higher total scores mean higher risk of losing the general oral health.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Median (Full Range); unit: Score on index
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
Score on index
  First assessment | 52 [46 to 52] | 52 [34 to 53]
  Last assessment | 52 [46 to 52] | 52 [34 to 53]

4. Primary Outcome: Change in Eating Assessment Tool (EAT-10)
Description: Swallowing quality of the patients will be assessed with eating assessment tool (EAT-10). the tool has ten questions and the total score of the tool is 40 points. Minimum score is 0 point and the maximum score is 40 point. Higher total scores mean higher risk of losing the general oral health.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
score on a scale
  First assessment | 0 [0 to 6] | 0 [0 to 5]
  Last assessment | 0 [0 to 4] | 0 [0 to 5]

5. Primary Outcome: Change in Pain Pressure Threshold of the Masticatory Muscles
Description: Two points in the masseter muscle and two points at the temporalis muscle, in total four points will be measured for the pain pressure threshold assessment. Measurements will be taken four times from every point with two-minute intervals. Due to first measurement values are generally high, average of the last three measurements will be calculated and recorded.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Median (Full Range); unit: kilogram
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
kilogram
  Right anterior temporalis first measurement | 2.3 [1.9 to 3.06] | 1.86 [1.56 to 2.56]
  Right anterior temporalis last measurement | 2.3 [2 to 2.76] | 1.86 [1.66 to 2.60]
  Left anterior temporalis first measurement | 2.3 [1.9 to 2.96] | 1.83 [1.6 to 2.5]
  Left anterior temporalis last measurement | 2.33 [2 to 2.66] | 1.8 [1.7 to 2.63]
  Right middle temporalis first measurement | 2.3 [2 to 3.16] | 1.91 [1.70 to 2.73]
  Right middle temporalis last measurement | 2.5 [2 to 2.86] | 1.95 [1.76 to 2.7]
  Left middle temporalis first measurement | 2.3 [2 to 3.13] | 1.9 [1.7 to 2.7]
  Left middle temporalis last measurement | 2.43 [2 to 2.83] | 1.9 [1.8 to 2.73]
  Right anterior masseter first measurement | 1.5 [1.36 to 1.86] | 1.3 [1.1 to 1.76]
  Right anterior masseter last measurement | 1.5 [1.2 to 1.66] | 1.3 [1.2 to 1.83]
  Left anterior masseter first measurement | 1.5 [1.13 to 1.83] | 1.3 [1.1 to 1.8]
  Left anterior masseter last measurement | 1.5 [1.1 to 1.66] | 1.31 [1.2 to 1.8]
  Right inferior masseter first measurement | 1.4 [1.3 to 1.8] | 1.24 [1.1 to 1.66]
  Right inferior masseter last measurement | 1.46 [1.1 to 1.73] | 1.3 [1.2 to 1.73]
  Left inferior masseter first measurement | 1.5 [1.13 to 1.7] | 1.2 [1.1 to 1.7]
  Left inferior masseter last measurement | 1.46 [1.1 to 1.6] | 1.3 [1.1 to 2.1]

6. Primary Outcome: Change in Craniocervical Angle Measurement
Description: Measurement will be taken while the patients are seated and their head in natural position. After that photos of the patients will be taken and then processus spinosus of the C7 and the tragus of the ear will be marked. After that, the angle between those to marking will be measured by the protractor.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
degree
  First measurement | 28.93 (12.54) | 29.09 (11.95)
  Last measurement | 27.07 (12.57) | 30.53 (11.95)

7. Primary Outcome: Change in Repeated Saliva Swallow Test
Description: Patients will be asked to swallow their saliva as much as they can do in thirty seconds.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Median (Full Range); unit: mililiter
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
mililiter
  First assessment | 3 [2 to 6] | 2.5 [2 to 4]
  Last assessment | 3 [2 to 6] | 3 [2 to 4]

8. Primary Outcome: Change in Fonseca Questionnaire
Description: Temporomandibular joint dysfunction existence and its severity will be assessed with Fonseca Questionnaire. Questionnaire includes 10 questions with yes, sometimes and no answers matching with 10, 5, and 0 point. Total score of the questionnaire is 100 point. Categorization of dysfunction by the questionnaire as follows; 70-100 point: severe dysfunction, 45-65: moderate dysfunction, 20-40: mild dysfunction and 0-15: has no dysfunction at all.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
score on a scale
  First value | 25 [20 to 40] | 20 [20 to 40]
  Last value | 25 [10 to 40] | 20 [15 to 30]

9. Primary Outcome: Change in Intraoral pH Measurement
Description: Saliva of the patients will be collected between 08:00-12:00 am. After the saliva collected in centrifuge tube reaches 5 ml, collection process will be stopped and immediately pH of the saliva measured with two decimal digital pH meter
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
pH
  First measurement | 6.45 (0.28) | 6.66 (0.4)
  Last measurement | 6.54 (0.3) | 6.63 (0.34)

10. Primary Outcome: Change in Neck Flexor Endurance Test
Description: Test will be performed while the patients are in supine position. After the position is taken patient will be asked to elevate their head about one inch and keep it that way as much as they can do. The period that passes from starting to the positional alteration will be recorded as the test score.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
second
  First assessment | 24.02 (10.89) | 27.12 (11.58)
  Last assessment | 26.97 (14.25) | 27.92 (10.58)

11. Secondary Outcome: Mini Mental State Exame Test
Description: Mini mental state exam test that consist of eleven articles will be used to assess whether the patients' mental state meets for the study enrollment. Total score is maximum 30 point. Lower score characterized with cognitive dysfunction. Cut off point of the test is 24 point or higher which means no cognitive impairment. 18 to 23 point means mild cognitive dysfunction. Total score below the 18 point means severe cognitive dusfunction. Minimum score is zero maximum score is 30.
Time Frame: At the enrollment process
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
score on a scale | 26.13 (1.73) | 25.06 (0.93)

12. Secondary Outcome: Change in Labial Commissure Angle
Description: Facial asymmetry of the patients will be assessed with labial commissure angle measurements. Black and white photos of the patients will be taken while the patients are in a seating position. Then photo will be printed in A5 sheet. After that, the angle between bilateral labial commissures, glabella, and the mental protuberance will be measured. Reference value of the labial commissure angle is approximately 90 degrees.
Time Frame: Two measurements: At the beginning and after three weeks
Measure: Mean (Full Range); unit: degree
Arm/Group | Expiratory Muscle Training Group | Control Group
Number analyzed (Participants) | 15 | 16
degree
  First measurement | 91 [83.5 to 93] | 92 [89 to 98]
  Last measurement | 90 [85 to 92] | 90.5 [89 to 95]

ADVERSE EVENTS:
Time Frame: During the patient specific time frame which is 3 weeks no adverse event has occurred.
Groups:
- Expiratory Muscle Training Group: Consisted of stroke patients using the expiratory muscle training device.
- Control Group: Stroke patients that have enrolled to the hospital conventional physiotherapy program.
Arm/Group | Expiratory Muscle Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

LIMITATIONS AND CAVEATS:
Due to COVID-19 pandemic, portable maximum expiratory pressure measurement device couldn't be used for this reason expiratory muscle device was calibrated based on patients' subjective feedback.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04569968/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04569968/SAP_001.pdf
  • Informed Consent Form (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04569968/ICF_002.pdf